CLINICAL TRIAL: NCT04769115
Title: A Predictive Technology for Prevention of Diabetic Foot Ulcers, and in Real Time, Identifying Diabetic Patients Who Experience Lower Extremity Trauma and Vascular Obstruction Utilizing the Science of Temperature (Inflammation) Trending
Brief Title: A Predictive Technology for Prevention of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DAPS Health LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20204536
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Diabetics who have no history of lower extremity (LEX) complications Diabetics who a history of LEX complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Response to Alerts (Other): Monitor patients daily for response to temperature changes and provide referral to doctor as needed
  Interventions: Device: Alert for temperature delta

INTERVENTIONS:
Device: Alert for temperature delta — If alert for potential complications refer to appropriate specialist

SUMMARY:
The DAPSHealth system employs a predictive technology for prevention of diabetic foot ulcers, and in Real Time, identifies diabetic patients who experience lower extremity trauma and vascular obstruction utilizing the science of temperature trending.

DETAILED DESCRIPTION:
Diabetes has become a major health issue in the United States and globally, particularly among older populations. There are currently 400 million diabetics worldwide, with 30 million diagnosed diabetics living in the US.

The standard of care today in treating complications of diabetes is a reactive one: doctors often wait for a problem to occur and then treat it. This waiting approach results in high medical expenses and an increase in pain for patients.

This study is testing a predictive technology system (investigational bluetooth-enabled thermometer and mobile app) to see if it can identify potential foot complications before the damage becomes irreversible. The thermometer being used in this study is the Exergen DermaTemp (DT) Thermometer. Participants will check the temperature of each foot daily for a period of three months. These results will sync directly from the thermometer to the mobile app.

Patients are notified when temperature levels indicate a potential complication that may lead to a developing foot ulcer. The study doctor is available to determine if any trauma or vascular obstruction has occurred and will follow up with the participant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes
* ambulatory
* smart device

Exclusion Criteria:

* non-ambulatory
* no smart device

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Predicting diabetic foot complications | Evaluate results daily and compare previous results to analyze multiple days with a contralateral delta of 4 degrees or more. This will be a running comparison over the three months of the trial.
  Monitor patients daily for inflammatory responses to trauma to avoid complications.
  This examines multiple plantar points on each foot and does a contralateral comparison to ensure there is no inflammatory response equal or greater than 4 degrees F between each pair. When this occurs over multiple days, we alert the patient to contact their physician. The temperature readings will be recorded using the DAPS Health system comprised of the Exergen DermaTemp 2000 FootScanner, DAPS Health Application and backend analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sussman, Dr., Principal Investigator — DAPS Health LLC
Locations (1):
- Annapolis Foot & Ankle, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All temperature data analysis (Alerts and disposition) based on patient history
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of completion of study
Access Criteria: not yet determined